CLINICAL TRIAL: NCT07272538
Title: The Role of FRAIL and FIND Frailty Scales in Predicting Chemotherapy-Related Toxicity Among Older Adults Receiving Adjuvant Treatment for Gastrointestinal Cancers: A Prospective Observational Study
Brief Title: Predicting Chemotherapy Toxicity Using FRAIL and FIND in Older Adults With Gastrointestinal Cancers
Acronym: FRAIL-GI
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, MD, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-125; AEŞH-EK-2025-125 (Other: Clinical Research Ethics Committee of Ankara Etlik City Hospital)
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Cancers; Frailty at Older Adults; Chemotherapy
Keywords: Geriatric Oncology; Older Adults; Frailty; FRAIL Scale; FIND Questionnaire; Chemotherapy Toxicity; Adjuvant Chemotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant Chemotherapy Cohort: This cohort includes older adults (age ≥65 years) with resected gastrointestinal cancers who received standard adjuvant chemotherapy (FOLFOX, CAPEOX, or capecitabine). All participants underwent frailty assessments using the FRAIL and FiND instruments at baseline, mid-treatment, and end of treatment. No intervention was assigned. This group reflects real-world observational follow-up of 84 consecutively treated patients.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This study assigned no intervention. Participants received standard-of-care adjuvant chemotherapy according to routine clinical oncology practice. The study observed frailty assessments and toxicity outcomes only.

SUMMARY:
This observational study evaluated whether two frailty screening tools, the FRAIL scale and the FiND questionnaire, can predict chemotherapy-related side effects in older adults with gastrointestinal cancers. Patients aged 65 years or older who received standard adjuvant chemotherapy after curative surgery for cancers of the colon, rectum, stomach, pancreas, or esophagus were included. No experimental treatment was given, and all patients received routine chemotherapy determined by their treating oncologists.

Frailty was assessed at the beginning of chemotherapy, around the middle of treatment, and at the end of therapy. Side effects were recorded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The main goal was to determine whether baseline frailty scores were associated with severe (Grade 3 or higher) chemotherapy toxicity. Additional goals included understanding how nutritional status, performance status, and comorbidities were related to toxicity and treatment completion.

The study collected real-world data to help identify older patients at higher risk of toxicity and to support safer, more personalized decision-making in routine oncology practice.

DETAILED DESCRIPTION:
This prospective observational study evaluated the relationship between frailty and chemotherapy-related toxicity in older adults with gastrointestinal cancers. Frailty was assessed using two validated screening tools: the FRAIL scale and the FiND questionnaire. Both tools are short, patient-reported screening instruments designed to identify vulnerability, reduced physiological reserve, and early mobility limitations in older adults. Both frailty instruments (FRAIL and FiND) have validated Turkish-language versions, ensuring cultural and linguistic appropriateness for use in older adults in Turkey.

Frailty Assessment Instruments

1. FRAIL Scale (Score Range: 0-5)

The FRAIL scale includes five items (Fatigue, Resistance, Ambulation, Illness, and Loss of weight).

Each item scores 1 point for "Yes" and 0 points for "No":

Fatigue: Feeling tired most or all of the time

Resistance: Difficulty climbing 10 steps

Ambulation: Difficulty walking one block

Illness: Having ≥5 chronic illnesses

Loss of Weight: Unintentional weight loss ≥5% in the past 6 months

Interpretation:

0 points: Robust

1-2 points: Pre-frail

3-5 points: Frail

2. FiND Questionnaire (Score Range: 0-5)

The FiND tool distinguishes frailty from mobility disability and includes five dichotomous questions:

Mobility Items:

Inability to walk 400 meters

Inability to climb one flight of stairs

Frailty Items:

Unintentional weight loss

Persistent fatigue

Reduction in physical activity

Interpretation:

0: Normal

1-2: Mild frailty or early disability

3-5: Frailty or mobility disability

Frailty assessments were conducted at baseline, mid-treatment (~3 months), and end of treatment (~6 months). Nutritional status was assessed with the Mini Nutritional Assessment-Short Form (MNA-SF), performance status with ECOG, and comorbidity burden with the modified Charlson Comorbidity Index (mCCI).

CTCAE v5.0 Toxicity Assessment

Chemotherapy-related adverse events were systematically recorded at each treatment cycle according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, focusing on clinically relevant toxicities frequently observed during fluoropyrimidine-based adjuvant chemotherapy.

Hematologic Toxicities

Neutropenia

Febrile neutropenia

Anemia

Thrombocytopenia

Gastrointestinal Toxicities

Nausea / vomiting

Diarrhea

Constipation

Mucositis / stomatitis

Neurologic Toxicities

Peripheral sensory neuropathy (oxaliplatin-related)

Constitutional Toxicities

Fatigue

Weight loss

Decreased appetite

Dermatologic Toxicities

Hand-foot syndrome (capecitabine-related)

Rash

Laboratory Abnormalities

Elevated liver enzymes

Renal function changes

Toxicity Grading

Toxicities were graded on a 5-point scale:

Grade 1-2: Mild to moderate

Grade 3: Severe, medically significant

Grade 4: Life-threatening

Grade 5: Treatment-related death

The primary endpoint was the incidence of Grade ≥3 toxicity. Secondary analyses explored dose delays, treatment reductions, early discontinuation, and associations between frailty dynamics and toxicity patterns.

Study Objective and Rationale

The study aimed to determine whether short, rapid frailty screens can help predict chemotherapy tolerance in older adults. Identifying patients at higher risk of toxicity may allow clinicians to personalize treatment intensity, optimize supportive care, and avoid unnecessary harm.

This research contributes real-world evidence supporting the integration of frailty screening into routine oncology practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Histologically confirmed gastrointestinal (GI) malignancy, including: Colorectal adenocarcinoma (colon or rectum), Gastric adenocarcinoma, Pancreatic adenocarcinoma, Biliary tract cancer (cholangiocarcinoma, gallbladder cancer) Small intestine adenocarcinoma, Esophageal cancer (adenocarcinoma or squamous cell carcinoma)
* Completion of curative-intent surgery with a postoperative plan for adjuvant chemotherapy.
* Receipt of standard adjuvant chemotherapy, including (but not limited to): FOLFOX, CAPOX (XELOX), Capecitabine monotherapy, FOLFIRINOX (selected fit older adults only), Gemcitabine ± capecitabine
* Initiation of adjuvant chemotherapy within the study period.
* Baseline frailty assessment (FRAIL Scale and FiND questionnaire) completed before the first chemotherapy cycle.
* Ability to provide informed consent and comply with frailty and toxicity follow-up assessments.

Exclusion Criteria:

* Age <65 years.
* Metastatic, recurrent, or unresectable disease at the time of adjuvant treatment.
* Receiving neoadjuvant-only treatment without subsequent adjuvant chemotherapy.
* Non-adenocarcinoma GI malignancies treated with protocols outside standard adjuvant chemotherapy (e.g., GIST receiving adjuvant imatinib; neuroendocrine tumors).
* Prior chemotherapy within 12 months for another malignancy.
* Missing baseline frailty assessment (FRAIL or FiND).
* Missing toxicity follow-up after chemotherapy initiation.
* Severe cognitive impairment, advanced dementia, or psychiatric illness preventing reliable questionnaire completion.
* Concurrent participation in another interventional clinical trial that may alter chemotherapy toxicity or functional outcomes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study included older adults (≥65 years) with gastrointestinal cancers who underwent curative-intent surgery and received standard adjuvant chemotherapy at Ankara Etlik City Hospital. A total of 84 participants were evaluated. All participants completed baseline frailty assessments (FRAIL and FiND) before chemotherapy initiation and were followed throughout the full adjuvant treatment course.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Association Between Baseline Frailty Scores (FRAIL and FiND) and the Incidence of Grade ≥3 Chemotherapy-Related Toxicity | From baseline (before the first chemotherapy cycle) through every chemotherapy cycle during the adjuvant regimen, with summary toxicity assessments performed at mid-treatment (~3 months) and at treatment completion (~6 months).
  This outcome examines whether baseline frailty, analyzed separately using the FRAIL Scale and the FiND Questionnaire, is associated with the development of severe chemotherapy-related toxicity. Toxicities were classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, where Grade 3 = severe, Grade 4 = life-threatening, and Grade 5 = death.
  Frailty Instruments:
  FRAIL Scale (Fatigue, Resistance, Ambulation, Illness, Loss of Weight): score range 0-5; higher scores indicate worse frailty.
  FiND Questionnaire (Frailty and Mobility Disability): score range 0-5; higher scores indicate worse frailty or mobility disability.
  Each frailty score will be analyzed independently for its association with severe chemotherapy-related toxicity.

SECONDARY OUTCOMES:
Change in FRAIL (Fatigue, Resistance, Ambulation, Illness, Loss of Weight) Scale Score Over Time | Baseline, 3 months, and 6 months.
  The FRAIL Scale ranges from 0 to 5 points, where higher scores indicate worse frailty. This outcome evaluates changes in FRAIL scores at baseline, mid-treatment (3 months), and end of treatment (6 months).
Change in FIND (Frailty and Mobility Disability) Questionnaire Score Over Time | Baseline, 3 months, and 6 months.
  The FiND Questionnaire ranges from 0 to 5 points, where higher scores indicate worse frailty or mobility disability. This outcome evaluates changes in FiND scores at baseline, 3 months, and 6 months.
Correlation Between FRAIL Scale and FIND Questionnaire Scores | Baseline, 3 months, and 6 months.
  This outcome evaluates correlations between the FRAIL Scale (0-5; higher = worse frailty) and the FiND Questionnaire (0-5; higher = frailty or mobility disability) at baseline, 3 months, and 6 months.
Change in Mini Nutritional Assessment-Short Form (MNA-SF) Score Over Time | Baseline, 3 months, and 6 months.
  The MNA-SF ranges from 0 to 14 points, where lower scores indicate worse nutritional status and higher malnutrition risk, whereas higher scores indicate better nutritional status. This outcome measures changes in MNA-SF scores across treatment.
Incidence of Chemotherapy-Related Toxicity Categories Classified by CTCAE Version 5.0 | From first chemotherapy cycle to end of treatment (~6 months).
  Chemotherapy-related toxicities were recorded at each cycle and classified using CTCAE v5.0 (Grade 1-5; higher grades indicate more severe toxicity). Categories include hematologic, gastrointestinal, neurologic, dermatologic, constitutional, and laboratory toxicities.
Association Between Changes in Frailty Scores and Development of Grade ≥3 Toxicity | Baseline to 6 months.
  This outcome evaluates whether increases in FRAIL score (0-5; higher = worse frailty) between baseline and follow-up (3 and 6 months) are associated with severe toxicity (Grade ≥3).
Proportion of Participants Completing All Planned Adjuvant Chemotherapy Cycles | End of planned adjuvant chemotherapy (~6 months).
  Completion is defined as receiving all planned cycles of adjuvant chemotherapy, regardless of dose modifications.
Incidence of Chemotherapy Treatment Modifications | From first chemotherapy cycle through the end of treatment (up to 6 months).
  Treatment modifications include any chemotherapy dose reduction, treatment delay, or permanent discontinuation due to toxicity. All modifications were prospectively recorded.
Correlation Between FRAIL Scale Score and Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline
  This outcome examines associations between the FRAIL Scale (0-5; higher = worse frailty) and the ECOG Performance Status (0-5; higher = worse functional capacity) at baseline.
Correlation Between FRAIL Scale Score and the Modified Charlson Comorbidity Index (mCCI) | Baseline
  This outcome evaluates the association between the FRAIL Scale score and comorbidity burden measured by the Modified Charlson Comorbidity Index (mCCI).
  FRAIL Scale range: 0-5 points; higher scores indicate worse frailty.
  mCCI has no fixed upper limit; higher scores indicate greater comorbidity burden.
  Correlation coefficients will be calculated to determine whether higher frailty scores are associated with higher comorbidity burden.
Predictive Performance of Baseline FRAIL Score for Grade ≥3 Toxicity | Baseline through 6 months.
  This outcome evaluates the ability of the FRAIL Scale score (0-5; higher = worse frailty) to discriminate between patients who do and do not develop severe toxicity (Grade ≥3), using receiver operating characteristic (ROC) curves and area under the curve (AUC) values.
Predictive Performance of Baseline FiND Score for Grade ≥3 Toxicity | Baseline through 6 months.
  This outcome evaluates the discriminative ability of the FiND Questionnaire score (0-5; higher = worse frailty or mobility disability) to identify patients who develop Grade ≥3 toxicity, using ROC curves and AUC values.
Association Between Changes in FIND Questionnaire Score and Development of Grade ≥3 Toxicity | Baseline to 6 months.
  This outcome evaluates whether worsening frailty or mobility limitation, defined as increases in FiND score (0-5), predicts Grade ≥3 chemotherapy-related toxicity.
Correlation Between FiND Questionnaire Score and Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline.
  This outcome evaluates correlations between the FiND score (0-5; higher = worse frailty or mobility disability) and ECOG status (0-5; higher = worse functional status).
Correlation Between FIND Questionnaire Score and the Modified Charlson Comorbidity Index (mCCI) | Baseline
  This outcome evaluates the association between the FiND Questionnaire score and comorbidity burden measured by the Modified Charlson Comorbidity Index (mCCI).
  FIND Questionnaire range: 0-5 points; higher scores indicate worse frailty or mobility disability.
  mCCI: higher scores indicate greater comorbidity burden.
  Correlation coefficients will be calculated to determine whether higher levels of frailty or mobility disability correlate with greater comorbidity burden.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital Medical Oncology Department, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes sensitive clinical information from older adults and cannot be fully de-identified without compromising data integrity. Data sharing is restricted by institutional ethics board regulations of Ankara Etlik City Hospital. Aggregated results will be made available upon publication.